CLINICAL TRIAL: NCT06083493
Title: Neuromodulation of Conscious Perception: Investigating Thalamic Roles Through Ultrasonic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zirui Huang, Research Assistant Professor, Anesthesiology and Research Fellow, Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00240514
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Thalamus
Keywords: Perception

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- LIFUP excitation (Experimental): The study will involve the enrollment of 60 participants, who will be randomly assigned to two groups, with each group consisting of 30 participants. The participants will be divided based on the type of transcranial LIFUP they will receive, either excitation or inhibition, targeting four specific thalamic areas.
  Interventions: Device: LIFUP excitation
- LIFUP inhibition (Experimental): The study will involve the enrollment of 60 participants, who will be randomly assigned to two groups, with each group consisting of 30 participants. The participants will be divided based on the type of transcranial LIFUP they will receive, either excitation or inhibition, targeting four specific thalamic areas.
  Interventions: Device: LIFUP inhibition

INTERVENTIONS:
Device: LIFUP excitation — The experimental will consist of a 10-minute baseline period (LIFUP-OFF) followed by four 10-minute sessions of stimulating (LIFUP-ON-excitation) four thalamic areas. The order of thalamic area stimulation will be counterbalanced across participants and will include the ventral anterior (VA), dorsal anterior (DA), ventral posterior (VP), and dorsal posterior (DP) sections of the thalamus.
  Arms: LIFUP excitation
Device: LIFUP inhibition — The experimental will consist of a 10-minute baseline period (LIFUP-OFF) followed by four 10-minute sessions of stimulating (LIFUP-ON-inhibition) four thalamic areas. The order of thalamic area stimulation will be counterbalanced across participants and will include the ventral anterior (VA), dorsal anterior (DA), ventral posterior (VP), and dorsal posterior (DP) sections of the thalamus.
  Arms: LIFUP inhibition

SUMMARY:
The purpose of this study is to evaluate the role that the thalamus (the egg-shaped structure in the middle of your brain) plays in perception using a low-intensity ultrasound pulsation (LIFUP) device. The researchers expect to observe differential changes in the perceptual outcomes based on the LIFUP stimulation of different thalamic areas

ELIGIBILITY:
Inclusion Criteria:

* Must be right-handed.
* Must have normal or corrected-to-normal vision (while wearing contact lenses). Please note: persons who need eyeglasses to achieve 20/20 vision cannot be included in this study as eyeglasses cannot be worn during the study visit.
* Must not be on any medications for any neurological, psychological, or psychiatric conditions.
* Must be English speaking.
* Must be capable of giving written informed consent.

Exclusion Criteria:

• Vision that is not 20/20, or vision that is not corrected to 20/20 while wearing contact lenses.

Please note: persons needing eyeglasses to achieve 20/20 vision cannot be included in this study as eyeglasses cannot be worn during the study visit.

* History of significant head injury with loss of consciousness.
* Learning disability or other developmental disorder.
* Medication use for any neurological, psychological, or psychiatric conditions.
* Any impairment (sensory or motor loss), activity, or situation that in the judgment of the study coordinator or Principal Investigators would prevent satisfactory completion of the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zirui Huang, Principal Investigator — University of Michigan; Anthony Hudetz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 participants were consented for this trial. 1 participant was excluded before randomization because of a scheduling conflict.
Period: Overall Study
Arm/Group | LIFUP Excitation | LIFUP Inhibition
Started | 30 | 30
Completed | 27 | 27
Not Completed | 3 | 3
Not completed — Technical issues with the interventional device | 2 | 2
Not completed — Performed incorrect visual task | 1 | 0
Not completed — Insufficient baseline performance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 61 participants consented, baseline data was not collected from 1 participant who was not randomized and did not participate in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | LIFUP Excitation | LIFUP Inhibition | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (7.0) | 24.5 (5.3) | 25.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7 | 9 | 16
  White | 20 | 19 | 39
  Black | 2 | 2 | 4
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Sensitivity Derived From the Signal Detection Theory (SDT)
Description: SDT was a means of measuring participants' ability to differentiate between information-bearing patterns and random patterns that distract from the information. Sensitivity measured a participant's ability to differentiate between real and scrambled images on a scale from 0.0 to 1.0, with higher scores indicating better accuracy in detecting a signal when it was present and lower scores indicating more missed signals. A score of 1.0 was perfect sensitivity (i.e., never missing a real signal).
Time Frame: Up to 60 minutes after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LIFUP Excitation | LIFUP Inhibition
Number analyzed (Participants) | 27 | 27
units on a scale
  Baseline | 0.7452 (0.1128) | 0.7419 (0.1250)
  Following intervention | 0.7520 (0.1014) | 0.7120 (0.1674)
Statistical Analysis 1: Comparison: LIFUP Excitation vs LIFUP Inhibition; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Perceptual Criterion Derived From the Signal Detection Theory (SDT)
Description: SDT was a means of measuring participants' ability to differentiate between information-bearing patterns and random patterns that distract from the information. Perceptual criterion measured a participant's tendency to say "yes" or "no" when the participant was unsure if a signal was present. Perceptual criterion was measured on a scale from -1.0 to 1.0, with a score of 0 indicating no bias towards "yes" or "no". Negative scores meant a bias towards "yes" (more likely to say a signal was present), while positive scores meant a bias towards "no" (more likely to say a signal was absent).
Time Frame: Up to 60 minutes after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LIFUP Excitation | LIFUP Inhibition
Number analyzed (Participants) | 27 | 27
units on a scale
  Baseline | 0.3008 (0.2589) | 0.2092 (0.2940)
  Following intervention | 0.3113 (0.3000) | 0.2770 (0.3322)
Statistical Analysis 1: Comparison: LIFUP Excitation vs LIFUP Inhibition; Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 32 days
Description: Adverse events were reviewed during the following 3 time points: at the time of the one-study visit, 24 hours via telephone after the study visit, and 30-days via medical chart review.
Arm/Group | LIFUP Excitation | LIFUP Inhibition
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIFUP Excitation (N=30) | LIFUP Inhibition (N=30)
Headache (Nervous system disorders) | 4 | 1
Fatigue (General disorders) | 1 | 0
Skin Irritation - Ear (Skin and subcutaneous tissue disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Dizziness (Ear and labyrinth disorders) | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Blurred Vision (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT06083493/Prot_SAP_000.pdf